CLINICAL TRIAL: NCT01666080
Title: Second or Greater Allogeneic Hematopoietic Stem Cell Transplant Using Reduced Intensity Conditioning (RIC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012OC065; MT2012-11C (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2012-07-31; First posted 2012-08-16 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hematologic Disorders; Hemoglobinopathies; Immunodeficiencies
Keywords: second stem cell transplant; donor hematopoietic engraftment; hematopoietic stem cell transplantation; inherited metabolic disorder
MeSH Terms: conditions — Hematologic Diseases; Hemoglobinopathies; Immunologic Deficiency Syndromes | interventions — Busulfan; fludarabine; fludarabine phosphate; Whole-Body Irradiation; Stem Cell Transplantation; Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced Intensity Conditioning (Other): Includes patients receiving a second or greater allogeneic hematopoietic stem cell transplant (HSCT) using reduced intensity conditioning (RIC). Patients will receive busulfan, fludarabine, total body irradiation and stem cell transplant. Keppra will be given for seizure prophylaxis.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Radiation: Total body irradiation; Biological: Stem cell transplant; Drug: Keppra

INTERVENTIONS:
Drug: Busulfan — 0.4 mg/kg (0.5 mg/kg if <4 years of age) intravenously (IV) every 6 hours on Days -8 and -7.
  Other Names: Busulfex
Drug: Fludarabine — 40 mg/m^2 intravenously (IV) over 1 hour on days -6 through -2.
  Other Names: Fludara
Radiation: Total body irradiation — 200 cGy on Day -1
Biological: Stem cell transplant — stem cell infusion on day 0
Drug: Keppra — Keppra will be given for seizure prophylaxis during busulfan administration as per the standard institutional protocol.
  Other Names: Levetiracetam

SUMMARY:
This is a treatment guideline for a second or greater allogeneic hematopoietic stem cell transplant (HSCT) using a reduced intensity conditioning (RIC) in patients with non-malignant or malignant diseases. This regimen, consisting of busulfan, fludarabine, and low dose total body irradiation (TBI), is designed to promote engraftment in patients who failed to achieve an acceptable level of donor-derived engraftment following a previous allogeneic HCT.

DETAILED DESCRIPTION:
There is no research element except the collection of routine clinical data. Patients will consent to allow routine clinical data to be collected and maintained in OnCore, the Masonic Cancer Center's (MCC) clinical database, and specific transplant related endpoints in the University Of Minnesota Blood and Bone Marrow Database as part of the historical database maintained by the department.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any disease for which a second or greater hematopoietic stem cell transplant is needed due to insufficient donor chimerism following hematopoietic recovery after previous HSCT. Determination of "insufficiency of donor chimerism" will be made by the treating transplant physician. Occasionally donor derived engraftment may be present, but sustained aplasia or failed recovery of sufficient hematopoiesis requires administration of a second graft. This intervention may be used for both situations.
* Donor Availability: Patients considered for transplantation must have a sufficient graft as based on current criteria of the University of Minnesota Blood and Marrow Transplantation Program

  * Transplantation using sufficiently matched related donors (such as matched siblings) or unrelated donors will be considered. Both granulocyte-colony stimulating factor (GCSF) stimulated peripheral blood grafts and bone marrow grafts will be considered, although bone marrow will be the priority.
  * Cord blood grafts, both related and unrelated, are also eligible. As this protocol will use a reduced intensity regimen, this protocol will use the current recommendations of the University of Minnesota for choosing cord blood grafts. If a single cord blood unit cell dose is insufficient, double cord transplantation should be considered if sufficiently matched cord blood units are available. The priority of choosing cord blood donors is based on the current institutional recommendations.
  * Exclusion of Metabolic Disorder or other Inherited Disorder Carrier Status from related donor and unrelated cord blood grafts as appropriate for primary disease.

At the discretion of the treating transplant physician, an allograft from the previous donor may be used, if available.

* Age, Performance Status, Consent

  * Age: 0 to 55 years
  * Consent: voluntary written consent (adult or parental/guardian)

Exclusion Criteria:

* Previous irradiation that precludes the safe administration of an additional dose of 200 cGy of total body irradiation (TBI). Radiation Oncology will evaluate all patients who have had previous radiation therapy or TBI for approval to receive an additional 200 cGy of TBI
* Pregnant or breastfeeding
* Active, uncontrolled infection - infection that is stable or improving after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections) will be permitted
* HIV positive
* While it would be advantageous to begin therapy on this second transplant regimen > 6 months following a prior myeloablative regimen or >2 months after a reduced intensity regimen, it is recognized that there are circumstances where this may not be practical.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Time to Engraftment | Day 42
  Neutrophil engraftment is defined as the first day of three consecutive days where the neutrophil count (absolute neutrophil count) is 500 cells/mm3 (0.5 x 109/L) or greater.

SECONDARY OUTCOMES:
Incidence of Graft Failure | Day 42
  Graft failure is defined as not accepting donated cells. The donated cells do not make the new white blood cells, red blood cells and platelets.
Status of Donor Chimerism | Day 100, 6 Months, 1 Year
  A state in bone marrow transplantation in which donor hematopoietic cells and host cells exist compatibly without signs of rejection.
Incidence of Acute Graft-Versus-Host Disease (GVHD) | Day 100
  Acute Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host.
Change in Incidence of Chronic Graft-Versus-Host Disease (GVHD) | 6 Months, 1 Year
  Chronic Graft-Versus-Host Disease is a severe long-term complication created by infusion of donor cells into a foreign host.
Incidence of Transplant Related Mortality | 6 Months
  In the field of transplantation, toxicity is high and all deaths without previous relapse or progression are usually considered as related to transplantation.
Incidence of Overall Survival | 6 Months
  The percentage of people in a study or treatment group who are alive for a certain period of time after they were diagnosed with or treated for a disease. Also called survival rate.
  Overall survival will be defined as time from date of enrollment to date of death or censored at the date of last documented contact for patients still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Troy Lund, M.D., Ph.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States